CLINICAL TRIAL: NCT02943993
Title: Non-Interventional Study on Edoxaban Treatment in Routine Clinical Practice in Patients With Venous Thromboembolism in Europe
Brief Title: Edoxaban Treatment in Routine Clinical Practice in Patients With Venous Thromboembolism in Europe
Acronym: ETNA-VTE
Status: Completed | Type: Observational
Sponsor: Daiichi Sankyo Europe, GmbH, a Daiichi Sankyo Company (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Other Study IDs: DSE-EDO-05-14-EU
Record Dates: First submitted 2016-10-24; First posted 2016-10-25 (Estimated); Results first posted 2022-05-02 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Venous Thromboembolism
Keywords: Post-Authorisation Safety Study; Real World Evidence; Edoxaban; Efficacy/Safety
MeSH Terms: conditions — Venous Thromboembolism | interventions — edoxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients treated with Edoxaban: Patients with established initial or recurrent acute symptomatic VTE treated with edoxaban according to the Summary of Product Characteristics (SmPC). Physician's prescribing behaviour will not be influenced, patients may only be included after the treating physician has made the clinical decision to prescribe edoxaban.
  Interventions: Drug: Edoxaban

INTERVENTIONS:
Drug: Edoxaban — Prescribed according to approved label
  Other Names: Lixiana

SUMMARY:
According to current guidelines, duration of anticoagulant treatment after a venous thromboembolic event varies from 3 months to indefinite treatment depending on the estimated risks of venous thromboembolism (VTE) recurrence and bleeding. Current data for edoxaban are limited to a maximum treatment duration of 12 months (Hokusai-VTE; N Engl J Med. 2013; 369:1406-15).

Therefore, this study aims to gather further insight into efficacy (i.e. symptomatic recurrent VTE) and safety (i.e. bleeding events, liver adverse events, all-cause mortality and other drug related adverse events) of extended treatment with edoxaban up to 18 months in an unselected patient population in routine clinical practice.

DETAILED DESCRIPTION:
Real-world evidence data in routine clinical practice use of edoxaban up to 18 months will be collected in 2,700 patients, treated by specialized as well as non-specialized physicians in hospitals and office based centres in 8 European countries. Patients from different countries and care settings (primary care and secondary care, different specialties) will be enrolled in this post-authorization safety study. Documentation of baseline and follow up information at 1, 3, 6, 12, and 18 months (only when available) will be collected. In addition, recurrence of symptomatic VTE and death will be captured retrospectively at time point of Last Patient Out per country.

Patients who discontinue permanently edoxaban during the observational period will be followed up according to the same scheme.

ELIGIBILITY:
Inclusion Criteria:

* Established acute initial or recurrent VTE
* Clinical decision for treatment with edoxaban is made at the time of enrollment
* Written informed consent for participation in the study (ICF)
* Not simultaneously participating in any interventional study

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with established initial or recurrent acute symptomatic VTE (distal or proximal deep vein thrombosis/pulmonary embolism) treated with edoxaban according to the Summary of Product Characteristics (SmPC). To ensure that the physician's prescribing behaviour will not be influenced, patients may only be included after the treating physician has made the clinical decision to prescribe edoxaban. Patients must have provided written informed consent for participation in the study (ICF) and should not participate simultaneously in any interventional study.
Sampling Method: Non-Probability Sample
Enrollment: 2809 (Actual)
Dates: Start 2016-04-06 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (1):
- International Clinical Research GmbH, Germering, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giugliano RP, Ruff CT, Braunwald E, Murphy SA, Wiviott SD, Halperin JL, Waldo AL, Ezekowitz MD, Weitz JI, Spinar J, Ruzyllo W, Ruda M, Koretsune Y, Betcher J, Shi M, Grip LT, Patel SP, Patel I, Hanyok JJ, Mercuri M, Antman EM; ENGAGE AF-TIMI 48 Investigators. Edoxaban versus warfarin in patients with atrial fibrillation. N Engl J Med. 2013 Nov 28;369(22):2093-104. doi: 10.1056/NEJMoa1310907. Epub 2013 Nov 19. PMID 24251359
- [Background] Hokusai-VTE Investigators; Buller HR, Decousus H, Grosso MA, Mercuri M, Middeldorp S, Prins MH, Raskob GE, Schellong SM, Schwocho L, Segers A, Shi M, Verhamme P, Wells P. Edoxaban versus warfarin for the treatment of symptomatic venous thromboembolism. N Engl J Med. 2013 Oct 10;369(15):1406-15. doi: 10.1056/NEJMoa1306638. Epub 2013 Aug 31. PMID 23991658
- [Derived] Cohen AT, Hoffmann U, Hainaut P, Gaine S, Ay C, Coppens M, Schindewolf M, Jimenez D, Bruggenjurgen B, Levy P, Laeis P, Fronk EM, Zierhut W, Malzer T, Manu MC, Reimitz PE, Bramlage P, Agnelli G; ETNA-VTE-Europe investigators. ETNA VTE Europe: A contemporary snapshot of patients treated with edoxaban in clinical practice across eight European countries. Eur J Intern Med. 2020 Dec;82:48-55. doi: 10.1016/j.ejim.2020.08.014. Epub 2020 Aug 18. PMID 32826158
- [Derived] Cohen AT, Ay C, Hainaut P, Decousus H, Hoffmann U, Gaine S, Coppens M, da Silva PM, Castro DJ, Amann-Vesti B, Bruggenjurgen B, Levy P, Bastida JL, Vicaut E, Laeis P, Fronk EM, Zierhut W, Malzer T, Bramlage P, Agnelli G; ETNA-VTE-Europe investigators. Design and rationale of the non-interventional, edoxaban treatment in routiNe clinical prActice in patients with venous ThromboEmbolism in Europe (ETNA-VTE-Europe) study. Thromb J. 2018 May 1;16:9. doi: 10.1186/s12959-018-0163-7. eCollection 2018. PMID 29719492

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 2809 participants were included in the All Documented Patient Set defined as participants with a signed ICF and trustworthy data at sites in Germany, Austria, Switzerland, Belgium, The Netherlands, United Kingdom, Ireland, and Italy; a total of 2655 participants were included in the Baseline Analysis Set and a total of 2644 participants were included in the Full Analysis Set.
Groups:
- ETNA-VTE: Participants with established initial or recurrent acute symptomatic venous thromboembolism (VTE) who were treated with edoxaban according to the Summary of Product Characteristics (SmPC) based on the clinical decision of the treating physician.
Period: Overall Study
Arm/Group | ETNA-VTE
Started | 2655 (Disposition data are based on Baseline Analysis Set (BAS) defined as All-Documented Patient Set participants with any documentation at the Baseline data collection point who fulfil the BAS criteria.)
Full Analysis Set | 2644
Completed | 2325
Not Completed | 330
Not completed — Withdrawal by Subject | 52
Not completed — Transfer to another institution | 6
Not completed — Lost to Follow-up | 135
Not completed — Death | 98
Not completed — Other reason for premature termination | 32
Not completed — Missing reason for termination | 7

BASELINE CHARACTERISTICS:
Population: Demographic and baseline characteristics were assessed in the Full Analysis Set.
Groups:
- ETNA-VTE: Participants with established acute initial or recurrent VTE who were treated with edoxaban according to Summary of Product Characteristics (SmPC) based on the clinical decision of the treating physician.
Arm/Group | ETNA-VTE
Number analyzed (Participants) | 2644
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 65.0 [52.0 to 76.0]
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 1312
  ≥65 and <75 years | 593
  ≥75 years | 739
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1231
  Male | 1413
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Germany | 722
  Austria | 182
  Switzerland | 84
  Belgium | 372
  Netherlands | 321
  United Kingdom | 113
  Ireland | 17
  Italy | 833

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With At Least 1 Symptomatic Venous Thromboembolism Recurrence - Overall
Description: Descriptive statistics were used to report the number of participants with at least 1 symptomatic VTE recurrence. Recurrent VTE events were based on adjudicated events.
  For the overall symptomatic VTE, precentage of participants (including 95% confidence intervals) were calculated.
Time Frame: Baseline up to end of observation period (18 months)
Population: VTE recurrence was assessed in the Full Analysis Set.
Measure: Number (95% Confidence Interval); unit: Percentage of VTE recurrence
Arm/Group | ETNA-VTE
Number analyzed (Participants) | 2644
Percentage of VTE recurrence | 3.8 [3.09 to 4.58]

2. Primary Outcome: Number of Participants With Bleeding Events (Adjudicated) While On Edoxaban Treatment
Description: Descriptive statistics were used to report the number of participants with bleeding events.
  For the analysis of bleeding events, absolute number of participants were calculated.
Time Frame: Baseline up to end of observation period (18 months)
Population: Bleeding events were assessed in the Full Analysis Set.
Measure: Number; unit: participants
Arm/Group | ETNA-VTE
Number analyzed (Participants) | 2644
participants
  Participants with any bleeding events | 304 [10.31 to 12.78]
  At least 1 major bleeding event | 38 [0.99 to 1.92]
  Clinically relevant non-major bleeding event | 82
  Minor | 300
  Gastrointestinal bleeding event | 77
  Epidural or subdural haematoma bleeding event | 4
  Intra-ocular bleeding event | 5
  Intra-articular bleeding event | 3
  Pleural bleeding event | 1
  Other bleeding event | 319
  Spontaneous bleeding | 287
  Provoked bleeding | 115
  Unknown bleeding | 18

3. Secondary Outcome: Percentage of Participants Experiencing At Least 1 Real World Safety Event - Overall
Description: Descriptive statistics were used to report the number of participants experiencing recurrent VTE and at least 1 real world safety event. VTE recurrence data were reported by recurrent deep vein thrombosis (DVT), recurrent pulmonary embolism (PE) with DVT, and recurrent PE only. Recurrent VTE events were based on adjudicated events. Real world safety events included all-cause death, cardiovascular (CV)-related death, VTE-related death, stroke, systemic embolic event, and hospitalization related to CV.
  For recurrent VTE and real world safety events, absolute and relative frequencies (including 95% confidence intervals) were calculated.
Time Frame: Baseline up to end of observation period (18 months)
Population: Real word safety events were assessed in the Full Analysis Set.
Measure: Number (95% Confidence Interval); unit: Percentage of real world safety events
Arm/Group | ETNA-VTE
Number analyzed (Participants) | 2644
Percentage of real world safety events
  Recurrent DVT only | 2.3 [1.77 to 2.95]
  Recurrent PE with DVT | 0.3 [0.11 to 0.54]
  Recurrent PE only | 1.2 [0.80 to 1.66]
  All-cause death | 3.6 [2.92 to 4.37]
  Cardiovascular-related death | 0.9 [0.55 to 1.30]
  Venous thromboembolism-related death | 0 [0 to 0.21]
  Stroke | 1.0 [0.64 to 1.44]
  Systemic embolic event | 0.1 [0.01 to 0.27]
  Hospitalization related to CV | 9.6 [8.47 to 10.75]

4. Secondary Outcome: Percentage of Participants With At Least 1 Symptomatic Venous Thromboembolism Recurrence - On Edoxaban Treatment
Description: Descriptive statistics were used to report the number of participants with overall symptomatic VTE recurrence. VTE recurrence data were further reported by recurrent deep venous thrombosis (DVT), recurrent pulmonary embolism (PE) with deep venous thrombosis (DVT), and recurrent PE only. Recurrent VTE events were based on adjudicated events.
  For symptomatic VTE recurrence, percentage of participants (95% confidence intervals) were calculated.
Time Frame: Baseline up to end of observation period (18 months)
Population: VTE recurrence was assessed in the Full Analysis Set.
Measure: Number (95% Confidence Interval); unit: Percentage of VTE recurrence
Arm/Group | ETNA-VTE
Number analyzed (Participants) | 2644
Percentage of VTE recurrence
  Recurrent VTE | 1.4 [0.99 to 1.92]
  Recurrent DVT only | 1.0 [0.67 to 1.48]
  Recurrent PE with DVT | 0 [0 to 0.21]
  Recurrent PE only | 0.3 [0.16 to 0.65]
  All-cause death | 1.9 [1.41 to 2.49]
  CV-related death | 0.4 [0.21 to 0.74]
  VTE-related death | 0 [0 to 0.21]
  Stroke | 0.6 [0.32 to 0.93]
  Systemic embolic event | 0 [0 to 0.21]
  Hospitalization-related to cardiovascular | 6.3 [5.42 to 7.31]

5. Secondary Outcome: Total Number of Venous Thromboembolism Recurrences By Type - Overall
Description: Descriptive statistics were used to describe the number of VTE events reported by the patient.
  For VTE recurrences, absolute number of VTE events were calculated.
Time Frame: Baseline up to end of observation period (18 months)
Population: Number of VTE recurrences were assessed in the Full Analysis Set.
Measure: Number; unit: VTE recurrences
Arm/Group | ETNA-VTE
Number analyzed (Participants) | 2644
VTE recurrences
  Total number of VTE recurrences | 105
  Deep vein thrombosis (DVT) only | 64
  Pulmonary embolism with DVT | 7
  Pulmonary embolism only | 32

6. Secondary Outcome: Duration of Venous Thromboembolism Recurrences, by Type - Overall
Description: Descriptive statistics were used to assess the duration of VTE events reported by the patient.
  For VTE recurrences, median duration of VTE events (interquartile range) were calculated.
Time Frame: Baseline up to end of observation period (18 months)
Population: Duration of VTE recurrences was assessed in patients with available start and stop data in the Full Analysis Set.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | ETNA-VTE
Number analyzed (Participants) | 2644
days
  Total number of VTE recurrences | 18.0 [8.0 to 93.0]
  Deep vein thrombosis (DVT) only | 44.5 [8.0 to 95.0]
  Pulmonary embolism with DVT | 8.0 [5.0 to 146.0]
  Pulmonary embolism only | 16.0 [8.0 to 93.0]

7. Secondary Outcome: Total Number of Venous Thromboembolism Recurrences (On Edoxaban Treatment)
Description: Descriptive statistics were used to assess the number of recurrent VTE events reported by the patient.
  For VTE recurrences, absolute number of VTE recurrences were calculated.
Time Frame: Baseline up to end of observation period (18 months)
Population: Number of VTE recurrences were assessed in the Full Analysis Set.
Measure: Number; unit: VTE recurrences
Arm/Group | ETNA-VTE
Number analyzed (Participants) | 2644
VTE recurrences
  Total number of VTE recurrences | 39
  Deep vein thrombosis (DVT) only | 28
  Pulmonary embolism with DVT | 1
  Pulmonary embolism only | 9

8. Secondary Outcome: Duration of Venous Thromboembolism Events (On Edoxaban Treatment)
Description: Descriptive statistics were used to assess the duration of VTE events reported by the patient.
  For VTE events, median duration of VTE events (interquartile range) were calculated.
Time Frame: Baseline up to end of observation period (18 months)
Population: Duration of VTE recurrences was assessed in patients with available start and stop data in the Full Analysis Set.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | ETNA-VTE
Number analyzed (Participants) | 2644
days
  Total number of VTE recurrences | 11.0 [8.0 to 20.0]
  Deep vein thrombosis (DVT) only | 9.5 [8.0 to 20]
  Pulmonary embolism with DVT | 0 [0 to 0]
  Pulmonary embolism only | 15.0 [8.0 to 16.0]

9. Secondary Outcome: Number of Participants With Risk Factors for Thromboembolic Events at Baseline
Description: Descriptive statistics were used to assess the number of participants with risk factors for thromboembolic events.
  For risk factors for thromboembolic events, absolute number of participants with risk factors (percentage) were calculated.
Time Frame: at Baseline
Population: Risk factors were assessed in the Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | ETNA-VTE
Number analyzed (Participants) | 2644
Participants
  Puerperium | 9
  Prolonged immobilisation | 401
  >5 days in bed | 218
  History of major surgery trauma | 359
  Known thrombophilic conditions | 111

10. Secondary Outcome: Duration of Edoxaban Treatment
Description: Descriptive statistics were used to report the duration of edoxaban treatment.
Time Frame: Baseline up to end of observational period (18 months)
Population: Duration of edoxaban treatment was assessed in the Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | ETNA-VTE
Number analyzed (Participants) | 2644
Participants
  Month 1 ongoing | 2527
  Month 3 ongoing | 2346
  Month 6 ongoing | 1842
  Month 12 ongoing | 1272
  Month 18 ongoing | 713
  Participants off edoxaban treatment at 18 months | 1910

11. Secondary Outcome: Number of Stroke Events
Description: Descriptive statistics were used to report the number of stroke events.
  For stroke events, absolute number of stroke events were calculated.
Time Frame: Baseline up to end of observation period (18 months)
Population: Stroke events were assessed in the Full Analysis Set.
Measure: Number; unit: events
Arm/Group | ETNA-VTE
Number analyzed (Participants) | 2644
events
  Overall treatment: Total number of stroke events | 27
  Overall treatment: Ischemic events | 17
  Overall treatment: Haemorrhagic events | 5
  Overall treatment: Unknown events | 5
  On treatment: Total number of stroke events | 16
  On treatment: Ischemic events | 12
  On treatment: Haemorrhagic events | 3
  On treatment: Unknown events | 1

12. Secondary Outcome: Number of Systemic Embolic Events - Overall
Description: Descriptive statistics were used to report the number of systemic embolic events (SEE).
  For SEE, absolute SEEs were calculated.
Time Frame: Baseline up to end of observation period (18 months)
Population: Systemic embolic events were assessed in the Full Analysis Set.
Measure: Number; unit: Systemic embolic events
Arm/Group | ETNA-VTE
Number analyzed (Participants) | 2644
Systemic embolic events
  Upper/lower extremity | 1
  Renal | 1

13. Secondary Outcome: Overview of Participants With Adverse Drug Reactions
Description: Descriptive statistics were used to report an overview of participants with adverse drug reactions (ADR). ADRs were coded using the Medical Dictionary for Regulatory Activities (MedDRA) version 20.1.
Time Frame: Baseline up to end of observation period (18 months)
Population: Adverse drug reactions were assessed in the Baseline Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | ETNA-VTE
Number analyzed (Participants) | 2655
Participants
  Death due to ADR | 2
  Participants with at least 1 ADR | 142
  Participants with at least 1 serious ADR | 59
  Study discontinuation due to ADR | 0

14. Secondary Outcome: Number of Participants With Adverse Drug Reactions by Preferred Term (≥0.2%)
Description: Adverse drug reactions were reported and coded using the Medical Dictionary for Regulatory Activities (MedDRA) version 20.1.
Time Frame: Baseline up to end of observational period (18 months)
Population: Adverse drug reactions were assessed in the Baseline Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | ETNA-VTE
Number analyzed (Participants) | 2655
Participants
  Haemorrhage | 35
  Gastrointestinal haemorrhage | 12
  Menorrhagia | 12
  Epistaxis | 11
  Fatigue | 8
  Nausea | 8
  Dizziness | 7
  Rash | 7
  Headache | 5
  Pruritus | 5

15. Secondary Outcome: Number of Participants With Pre-defined Adverse Drug Reactions
Description: Descriptive statistics were used to report the number of participants with pre-defined adverse drug reactions (ADR). ADRs were coded using the Medical Dictionary for Regulatory Activities (MedDRA) version 20.1.
Time Frame: Baseline up to end of observation period (18 months)
Population: Adverse drug reactions were assessed in the Baseline Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | ETNA-VTE
Number analyzed (Participants) | 2655
Participants
  Stroke | 2
  Bleeding events | 75
  Systemic embolic events | 0
  Non-valvular atrial fibrillation | 0
  Malignancy | 0
  Others | 4

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were not assessed in this non-interventional (observational) study.
Description: Treatment-emergent adverse events were not assessed in this non-interventional (observational) study. Adverse drug reactions were reported as a secondary outcome measure.
Arm/Group | ETNA-VTE
All-Cause Mortality (participants affected / at risk) | 98/2644
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-12): https://cdn.clinicaltrials.gov/large-docs/93/NCT02943993/Prot_SAP_000.pdf